CLINICAL TRIAL: NCT03727763
Title: Cetuximab and Vemurafenib Plus FOLFIRI for BRAF V600E Mutated Advanced Colorectal Cancer (IMPROVEMENT): A Single-arm Study
Brief Title: Cetuximab and Vemurafenib Plus FOLFIRI for BRAF V600E Mutated Advanced Colorectal Cancer (IMPROVEMENT)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Zhan Wang, A single center clinical study of FOLFIRI with vemurafenib and cetuximab in Advanced Colorectal Cancer Patients with BRAF V600E mutation., Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPROVEMENT
Record Dates: First submitted 2018-10-31; First posted 2018-11-01 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer
Keywords: FLOFIRI; vemurafenib; cetuximab; BRAF V600E mutation; Advanced Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Vemurafenib; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FIVC group (Experimental): Irinotecan 180mg/m2 iv gtt (14 days per course) leucovorin 400mg/m2 iv gtt (14 days per course) 5-fluorouracil 400mg/m2 iv (14 days per course) 5-fluorouracil 2400 mg/m2 46h (14 days per course) vemurafenib 960mg po bid cetuximab 500mg/m2 iv gtt (14 days per course)
  Interventions: Drug: Vemurafenib; Drug: Cetuximab

INTERVENTIONS:
Drug: Vemurafenib — 960mg po bid
  Other Names: PLX4032, RG7204
Drug: Cetuximab — 500mg/m2 iv gtt (14 days per course)
  Other Names: ERBITUX

SUMMARY:
This clinical trial aims to evaluate the efficacy, safety of FOLFIRI with vemurafenib and cetuximab in Advanced Colorectal Cancer Patients with BRAF V600E mutation.

ELIGIBILITY:
Inclusion Criteria:

* Patients have histologically or cytologically confirmed advanced or recurrent CRC;
* Patients with BRAV V600E mutation/KRAS WT based on the NGS or ARMS-PCR detection of tumor tissue;
* Patients have measurable disease as defined by RECIST 1.1 as determined by investigator;
* Patient with a history of radiotherapy at least 3 months before on the day of providing consent, but the measurable lesion should not be within the scope of radiotherapy;
* Patients without a history of receiving vemurafenib or cetuximab;
* Patients with age of 18-75yr;
* Patients with a performance status of 0,1or 2 on the Eastern Cooperative Oncology Group.；
* Patients with Life expectancy of more than 12 weeks;
* Patients must have the ability to understand and sign the written informed consent voluntarily;
* Female of childbearing potential who are negative in a pregnancy test within 14 days before enrollment. Both male and female patients should agree to use an adequate method of contraception (total abstinence, an intrauterine device or hormone releasing system, an contraceptive implant and an oral contraceptive) starting with the first dose of study therapy through 120 days after the last dose of study therapy. Duration will be determined when the subject is assigned to treatment.

Exclusion Criteria:

* Patients with KRAS/NRAS mutation;
* Patients with major surgery or severe trauma within 4 weeks before the first medication;
* Patients with hypersensitivity to the components in the study protocol;；
* Patients who are ready to give birth or are pregnant.。
* Patients with brain metastases 。
* Bone marrow, liver and kidney function did not meet the requirements of chemotherapy as follows：

  * Neutrophil count<1,500/mm3；
  * Platelet count <80,000/mm3；
  * Total bilirubin >1.5-times the upper limit of normal；
  * ALT/AST>2.5-times the upper limit of normal for patients without liver metastases; (5.0-times the upper limit of normal for patients without liver metastases)
  * Creatinine >1.5-times the upper limit of normal；
* Patients with cancers other than advanced colorectal cancer within five years prior to the start of treatment in this study. Cervical carcinoma in situ, cured basal cell carcinoma and bladder epithelial tumor were excluded;；
* Patients without legal capacity or limited civil capacity;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to 55 months
  Evaluation of tumor burden based on RECIST criteria every 3 cycles(each cycle is 14 days), ORR is the proportion of patients with reduction in tumor burden of a predefined amount, including complete response and partial response.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 55 months
  Evaluation of tumor burden based on RECIST criteria every 3 cycles(each cycle is 14 days), and DCR is the proportion of patients with reduction in tumor burden of a predefined amount, including complete response, partial response and stable disease
Progression-free survival | Time from treatment beginning until the date of first documented progression, assessed up to 55 months
  Evaluation of tumor burden based on RECIST criteria until first documented progress through study completion, an average of 6 weeks
Overall survival | Time from treatment beginning until date of death from any cause, assessed up to 55 months
  From date of treatment beginning until the date of death from any cause, through study completion, an average of 6 weeks
adverse events | Through study completion, an average of 4 weeks
  Incidence of Treatment-related adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Zhan Wang, Prof, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang Z, Qin BD, Ye CY, Wang MM, Yuan LY, Dai WP, Sun L, Liu K, Qin WX, Jiao XD, Li XN, Zang YS. Cetuximab and vemurafenib plus FOLFIRI (5-fluorouracil/leucovorin/irinotecan) for BRAF V600E-mutated advanced colorectal cancer (IMPROVEMENT): An open-label, single-arm, phase II trial. Eur J Cancer. 2022 Mar;163:152-162. doi: 10.1016/j.ejca.2021.12.028. Epub 2022 Jan 21. PMID 35074651